CLINICAL TRIAL: NCT03463551
Title: Perfluorocarbon (ABL-101) Oxygenation for Stroke: Trial With GOLD (Glasgow Oxygen Level Dependent Technology) Imaging Theranostic (POST-IT)
Brief Title: Perfluorocarbon (ABL-101) Oxygenation for Stroke: Trial With GOLD (Glasgow Oxygen Level Dependent Technology) Imaging Theranostic
Acronym: POST-IT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); Aurum Biosciences Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN16ST187
Record Dates: First submitted 2018-03-06; First posted 2018-03-13 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Acute Ischaemic Stroke
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABL-101 IV as per dosing cohort + Supplementary O2 for 24h (Experimental): Patients will receive either ABL-101 or placebo (equivalent volume of 0.9% Sodium Chloride) within ascending dose groups of 6 patients each (4 to ABL-101, 2 to placebo).The starting cohort will be Cohort 1: 0.5mL/kg.
  In the event that the start dose of Cohort 1 is considered intolerable in the opinion of the iDMC based on incidence of patients experiencing dose-limiting toxicities (DLTs), the iDMC will have the option of recommending a lower dose cohort (Cohort -1) of 0.25ml/kg (to a maximum of 25ml) be undertaken.
  Cohort 1: 0.5 mL/kg to a maximum of 50ml; Cohort 2: 1.5mL/kg to a maximum of 150ml; Cohort 3: 3.0mL/kg to a maximum of 300ml.
  All patients will receive Oxygen 60% by face mask (8l/min) for approximately 24h after ABL-101 or placebo administration.
  Interventions: Drug: ABL-101
- IV 0.9% NaCl as per dosing cohort + supplementary O2 for 24h (Placebo Comparator): Cohort 1: Volume matched to the calculation used for ABL-101 using patient weight; Cohort 2: Volume matched to the calculation used for ABL-101 using patient weight; Cohort 3: Volume matched to the calculation used for ABL-101 using patient weight.
  All patients will receive Oxygen 60% by face mask (8l/min) for approximately 24h after ABL-101 or placebo administration.
  Interventions: Other: 0.9% NaCl

INTERVENTIONS:
Drug: ABL-101 — ABL-101 is provided as a sterile phospholipid-based emulsion for intravenous administration.
  Arms: ABL-101 IV as per dosing cohort + Supplementary O2 for 24h
Other: 0.9% NaCl — Placebo
  Arms: IV 0.9% NaCl as per dosing cohort + supplementary O2 for 24h

SUMMARY:
This study evaluates the safety and tolerability of 3 dose levels of ABL-101 and supplemental oxygen in acute stroke patients.

DETAILED DESCRIPTION:
Only a small proportion of patients are currently suitable for treatment with "clot busting" drugs after a stroke. Being able to visualise potentially rescuable brain tissue on scanning may allow more people to be treated. Currently available methods require extra time to acquire and are not therefore widely used. By carrying significant extra oxygen to the brain, the ABL-101 molecule may not only allow the visualisation of salvageable tissue, but also prevent progression of stroke damage in and have an additional direct benefit on tissue survival. Studies in animal models of stroke show smaller areas of stroke damage after ABL-101. There is therefore a rationale for testing this molecule in stroke patients, both as a diagnostic method, and also as a potential therapeutic agent.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years.
* Males or females not of child-bearing potential defined as being post-menopausal based on cessation of regular menses for a minimum of 12 consecutive months with no alternative cause, permanently sterilised (e.g. hysterectomy, bilateral tubal occlusion, bilateral salpingectomy), or having medically confirmed ovarian failure.
* Ischaemic stroke <72h after onset.
* Previous functional independence (estimated mRS <3).
* Capacity to consent.

Exclusion Criteria:

* Women of child bearing potential.
* Contraindications to MRI scanning (eg cardiac pacemaker, ferromagnetic implants, known hypersensitivity to gadolinium containing contrast media).
* Known allergy to ABL-101 or any of its constituents, (including egg phospholipids).
* Clinical need for, or contraindication to, supplemental oxygen.
* Known impaired renal function (eGFR <30ml/min) precluding radiological contrast.
* Known thrombocytopaenia (platelet count <150x109) or history of platelet function disorder.
* Known intercurrent infection.
* Known severe COPD or cardiac failure (eg significantly limiting exercise capacity or requiring hospitalisation within the preceding 12 months).
* Known significant liver disease (eg liver failure or cirrhosis, chronic infectious or autoimmune hepatitis, or transaminases >3 times upper limit of normal).
* Any current medical condition causing impaired immunity (eg HIV infection, hyposplenism) or use of systemic immunosuppressant medication except for inhaled, nasal intra-articular or topical corticosteroids) on an ongoing basis or within the preceding 30 days.
* Any medical condition potentially limiting survival within the study follow-up period.
* Participation in another CTIMP within preceding 90 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of 3 dose levels of ABL-101 and supplemental oxygen in acute stroke patients. | 7 days±2
  Incidence of Serious Adverse Events and AEs of special interest up to visit 6 (day 7±2).

SECONDARY OUTCOMES:
Mortality | 30 days
Incidence of serious adverse events throughout the entire study period. | 30 days±5
Incidence of adverse events of special interest | 30 days±5
Incidence of adverse reactions, adverse events, serious adverse events and serious adverse reactions, up to visit 7 (30±5 days) post administration of Investigational medicinal product. | 30 days±5
Modified Rankin Scale (mRS) distribution at day 30. | At day 30
  The mRS is a hierarchical ordinal scale used to assess disability in stroke trials, with seven discrete levels that range from No Symptoms (mRS=0) to death (mRS=6). The Rankin Focused Assessment tool will be used to derive day 30 mRS.
Follow-up infarct volume on MRI brain at visit 4. | 48hrs (40-72hrs)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Muir, Principal Investigator — University of Glasgow

IPD SHARING:
Plan to Share IPD: No